CLINICAL TRIAL: NCT01662024
Title: Primary Obesity Multicenter Incisionless Suturing Evaluation: The PROMISE Trial
Brief Title: Endoscopic Suturing for Primary Obesity Treatment
Acronym: PROMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Thompson, Director of Therapeutic Endoscopy, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P-000799
Record Dates: First submitted 2012-06-15; First posted 2012-08-10 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Obesity; Body Weight; Overweight
Keywords: Obesity; BMI; Weight loss; Gastric restriction; Bariatrics
MeSH Terms: conditions — Obesity; Body Weight; Overweight; Weight Loss

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Endoscopic gastric restrictive procedure (Experimental): Restrict gastric size by approximating tissue endolumenally via an incisionless/per-oral approach.
  Interventions: Device: Endoscopic gastric restrictive procedure

INTERVENTIONS:
Device: Endoscopic gastric restrictive procedure — Endoluminal gastric tissue approximation using an incisionless/per-oral endoscopic suturing device for primary gastric restrictive procedures
  Other Names: Apollo Overstitch Endoscopic Suturing System

SUMMARY:
Gastric restriction is an important principle of both roux-en-Y gastric bypass and laparoscopic adjustable gastric banding. The FDA cleared OverStitch Endoscopic Suturing System (Apollo Endosurgery, Austin, TX) offers the physician the ability to restrict gastric size by approximating tissue endoluminally via an incisionless/per-oral approach. The use of this system has the potential to reduce the complications associated with current surgical approaches while effecting the desired gastric restriction. The primary objective is to collect data on the use of the OverStitch Endoscopic Suturing System (Apollo Endosurgery, Inc. Austin, Texas) for gastric tissue approximation during primary gastric restrictive procedures.

DETAILED DESCRIPTION:
The primary objective is to collect data on the use of the OverStitch Endoscopic Suturing System (Apollo Endosurgery, Inc. Austin, Texas) for gastric tissue approximation during primary gastric restrictive procedures.

The primary endpoint of this study is evaluation of safety and feasibility of the procedure. All subjects for whom the plication procedure is initiated (defined as placement of the overtube) will be included in the safety analysis. The primary safety analysis will assess the occurrence of adverse events through 12 months after the plication procedure.

Technical success will be defined as minimum placement of 8 sutures upon initial endoscopic intervention. Safety will be determined as no adverse events directly related to the procedure at 12 months.

Secondary Endpoints:

1. Efficacy: Data for the following effectiveness outcome measures (variables) will be collected and analyzed relative to baseline:

   * Percent excess weight loss (%EWL)
   * Total weight lost (kg) and percent weight lost
   * Change in (BMI) and percent change in BMI
   * Change in waist circumference
   * Improvement in co-morbid disease(s) including, but not limited to, improvement in vital signs and/or laboratory values
   * Changes in quality of life measures as reported on Quality of Life questionnaire(s) (evaluated relative to baseline)
   * Changes in feelings of satiety measures as reported on the TFEQ-R18 (relative to baseline)
2. Durability: Data will be collected on the durability of the plications by evaluating the remaining plications at the 12 month endoscopy, compared to the number of plications placed at the time of procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject has met diabetic lab testing and all pre-procedural qualifications
* Subject is ≥ 18 yrs. of age and ≤ 60 yrs. of age
* Subject has a BMI of > 30 and < 35
* Subject has history of obesity for > 2 yrs
* Subject has had no significant weight change (<5% of total body weight)in last 6 months
* Subject must have failed standard obesity therapy of diet, exercise, behavior modification, and pharmacologic agents either alone or in combination, as assessed by an interview with a member of the study team at baseline
* Subject is a reasonable candidate for general anesthesia
* Subject agrees not to have any additional weight loss surgery or reconstructive surgery that may affect body weight (i.e. mammoplasty, liposuction, lipoplasty, etc) during the trial
* Subject must be willing and able to participate in all aspects of the study and agree to comply with all study requirements for the duration of the study. This includes availability of reliable transportation and sufficient time to attend all follow-up visits.
* Subject must be able to fully understand and be willing to sign the informed consent

Exclusion Criteria:

* Subject has had significant weight loss in the last 3 months, or between baseline and the study procedure
* Mallampati (intubation) score greater than 3
* Subject is observed during EGD to have heavily scarred, malignant or poor quality/friable tissue in areas of the stomach where sutures are to be placed
* Subject has history or present use of insulin or insulin derivatives for treatment of diabetes
* Subject has diabetes secondary to a specific disease
* Subject has poorly controlled diabetes as indicated by the lack of stable diabetes medications and doses over the last month, or has a history of diabetes for greater than 10 years
* Subject has history of inflammatory disease of GI tract
* Subject has a history of intestinal strictures or adhesions
* Subject has renal and/or hepatic insufficiency
* Subject has chronic pancreatic disease
* Subject has history of/or signs and/or symptoms of gastro-duodenal ulcer disease and/or active peptic ulcer
* Subject has significant esophageal disease including Zenker's diverticulum, grade 3-4 reflux esophagitis, stricture, Barrett's esophagus, esophageal cancer, esophageal diverticulum, dysphagia, achalasia, or symptoms of dysmotility
* Subject has a history of any significant abdominal surgery
* Subject has had previous bariatric, gastric or esophageal surgery; intestinal obstruction; portal gastropathy; gastrointestinal tumors; esophageal or gastric varices, or gastroparesis
* Subject has a hiatal hernia > 2cm
* Subject has chronic/acute upper GI bleeding conditions
* Subject has severe coagulopathy (prothrombin time > 3 seconds over control or platelet count < 100,000) or is presently taking heparin, coumadin, warfarin, or other anticoagulants or other medications which impede coagulation or platelet aggregation
* Female subject is of childbearing age and not practicing effective birth control, is pregnant or is lactating
* Subject has symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
* Subject has cancer or life expectancy of < 2 yrs
* Subject has systemic infection in the body at the time of the plication procedure.
* Subject currently uses or has used over the counter or prescription weight loss medications in last 30 days or intends to use during follow-up Study period.
* Subjects who have started medications within the last 3 months that are known to cause weight gain
* Subjects undergoing chronic steroid therapy
* Subjects undergoing immunosuppressive therapy
* Subject has a history of drug or alcohol abuse
* Subject has a history of uncontrolled or poorly controlled psychiatric disease or suspected eating disorders
* Subject is non-ambulatory or has significant impairment of mobility
* Subject has known hormonal or genetic cause for obesity
* Subject is not in sufficient and stable medical health, as determined and evaluated by the Principal Investigator.
* Subject has participated in a clinical study with an investigational new drug, biological, or therapeutic device within ≤ 28 days prior to enrollment in this study, and does not agree to abstain from participation in other clinical trials of any kind during this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C. Thompson, MD, MS, Principal Investigator — Brigham and Women's Hospital
Locations (4):
- United States (4):
  - Jackson Health System, Miami, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - St. Joseph's Regional Medical Center at New Jersey, Paterson, New Jersey
  - University of Texas at Houston, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data is available immediately. We will share the outcomes data if a request is made via email to the PI and the data transfer is completed between institutions. Identifying information will not be provided.

REFERENCES:
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Willett WC, Dietz WH, Colditz GA. Guidelines for healthy weight. N Engl J Med. 1999 Aug 5;341(6):427-34. doi: 10.1056/NEJM199908053410607. No abstract available. PMID 10432328
- [Background] Dindo D, Muller MK, Weber M, Clavien PA. Obesity in general elective surgery. Lancet. 2003 Jun 14;361(9374):2032-5. doi: 10.1016/S0140-6736(03)13640-9. PMID 12814714
- [Background] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Background] Flum DR, Dellinger EP. Impact of gastric bypass operation on survival: a population-based analysis. J Am Coll Surg. 2004 Oct;199(4):543-51. doi: 10.1016/j.jamcollsurg.2004.06.014. PMID 15454136
- [Background] Szold A, Abu-Abeid S. Laparoscopic adjustable silicone gastric banding for morbid obesity: results and complications in 715 patients. Surg Endosc. 2002 Feb;16(2):230-3. doi: 10.1007/s004640080187. Epub 2001 Oct 5. PMID 11967669
- [Background] Jirapinyo P, Watson RR, Thompson CC. Use of a novel endoscopic suturing device to treat recalcitrant marginal ulceration (with video). Gastrointest Endosc. 2012 Aug;76(2):435-9. doi: 10.1016/j.gie.2012.03.681. Epub 2012 May 31. No abstract available. PMID 22658388

RESULTS

PARTICIPANT FLOW:
Groups:
- Endoscopic Gastric Restrictive Procedure: Restrict gastric size by approximating tissue endolumenally via an incisionless/per-oral approach.
  Endoscopic gastric restrictive procedure: Endoluminal gastric tissue approximation using an incisionless/per-oral endoscopic suturing device for primary gastric restrictive procedures. Dietitian visits were performed at 1, 3, 6, 9, and 12 months to assess for the development of eating disorders. Clinical visits were performed at 1, 3, 6, and 12 months to obtain size and weight data. Perioperative adverse events were defined as those occurring during the procedure or the post-procedure observation period.
Period: Overall Study
Arm/Group | Endoscopic Gastric Restrictive Procedure
Started | 20
Completed | 15
Not Completed | 5
Not completed — Pregnancy | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Adults who are suffering from obesity with a Body Mass Index (BMI) of 30 - 35 kg/m^2 seeking a minimally invasive alternative to bariatric surgery.
Arm/Group | Endoscopic Gastric Restrictive Procedure
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 36.7 [34.4 to 39.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Initial Weight (kg) [Mean (Full Range); unit: kg] | 90.4 [88.4 to 92.4]
Initial BMI (kg/m^2) [Mean (Full Range); unit: kg/m^2] | 33.4 [33.1 to 33.7]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Perioperative adverse events were defined as those occurring during the procedure or the post-procedure observation period. Postoperative adverse events were defined as occurring during the first three days after the procedure. Delayed adverse events were defined as occurring on the fourth post-procedure day or afterwards.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopic Gastric Restrictive Procedure
Number analyzed (Participants) | 20
Participants
  Peri-operative Adverse Events | 5
  Post-operative Adverse Events | 2
  Delayed Adverse Events | 0
  No Adverse Events | 13

2. Primary Outcome: Evaluation of Technical Feasibility of the Procedure
Description: Technical success was defined by placement of at least 8 running sutures and 4 interrupted sutures in the gastric body with exclusion of the lateral stomach.
Time Frame: Day 0 - Procedure Day
Measure: Mean (Full Range); unit: Sutures
Groups:
- Endoscopic Gastric Restrictive Procedure: Restrict gastric size by approximating tissue endolumenally via an incisionless/per-oral approach.
  Endoscopic gastric restrictive procedure: Endoluminal gastric tissue approximation using an incisionless/per-oral endoscopic suturing device for primary gastric restrictive procedures. D
Arm/Group | Endoscopic Gastric Restrictive Procedure
Number analyzed (Participants) | 20
Sutures
  Running Sutures | 10.4 [9.9 to 10.9]
  Total Stitches | 54.4 [51.9 to 56.9]
  Interrupted Sutures | 4 [4 to 4]

3. Secondary Outcome: Percent Excess Weight Loss
Description: Data for the following effectiveness outcome measures (variables) will be collected and analyzed relative to baseline: Percent excess weight loss
Time Frame: 12 Months
Measure: Mean (Full Range); unit: Percentage of excess weight lost
Arm/Group | Endoscopic Gastric Restrictive Procedure
Number analyzed (Participants) | 15
Percentage of excess weight lost | 70.8 [62.8 to 78.8]

4. Secondary Outcome: Durability
Description: Data will be collected on the durability of the plications by evaluating the remaining plications at the 12 month endoscopy, compared to the number of plications placed at the time of procedure.
Time Frame: 12 months
Population: Endoscopies were performed at 12 months but it was difficult to count the number of plications still intact as originally planned.
Arm/Group | Endoscopic Gastric Restrictive Procedure
Number analyzed (Participants) | 0
Value | 0

5. Secondary Outcome: Percentage of Total Body Weight Loss
Description: Data for the following effectiveness outcome measures (variables) will be collected and analyzed relative to baseline: Percentage of Total body weight loss
Time Frame: 12 Months
Measure: Mean (Full Range); unit: Percentage of total weight lost
Arm/Group | Endoscopic Gastric Restrictive Procedure
Number analyzed (Participants) | 15
Percentage of total weight lost | 18.1 [15.8 to 20.4]

6. Secondary Outcome: BMI Loss (kg/m^2)
Description: Data for the following effectiveness outcome measures (variables) will be collected and analyzed relative to baseline: BMI Loss (kg/m^2)
Time Frame: 12 Months
Measure: Mean (Full Range); unit: kg/m^2
Arm/Group | Endoscopic Gastric Restrictive Procedure
Number analyzed (Participants) | 15
kg/m^2 | 6.1 [5.3 to 6.9]

7. Secondary Outcome: Waist Circumference Loss (cm)
Description: Data for the following effectiveness outcome measures (variables) will be collected and analyzed relative to baseline: Waist Circumference Loss (cm)
Time Frame: 12 Months
Measure: Mean (Full Range); unit: cm
Arm/Group | Endoscopic Gastric Restrictive Procedure
Number analyzed (Participants) | 15
cm | 16 [13.6 to 18.4]

ADVERSE EVENTS:
Time Frame: 12 month period of adverse event data collection.
Arm/Group | Endoscopic Gastric Restrictive Procedure
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 7/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endoscopic Gastric Restrictive Procedure (N=20)
Perioperative Abdominal Pain (Gastrointestinal disorders) | 2 — Perioperative Adverse Event is on Day of procedure (Day 0)
Perioperative Nausea/Vomiting (Gastrointestinal disorders) | 3 — Perioperative Adverse Event is on Day of procedure (Day 0)
Post-operative Abdominal Pain (Gastrointestinal disorders) | 1 — Post-operative reporting is 1-3 days after the procedure
Post-operative Nausea (Gastrointestinal disorders) | 1 — Post-operative reporting is 1-3 days after the procedure

LIMITATIONS AND CAVEATS:
Early termination and withdrawal of 5 subjects leads to small numbers of subjects analyzed.

No sham comparator.

Durability measures at 12 month endoscopy was difficult to quantify.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No